CLINICAL TRIAL: NCT03653546
Title: A Randomized, Open-label, Controlled, Multi-Center Phase II/III Study to Assess the Efficacy and Safety of AZD3759 vs. a Standard of Care EGFR TKI, as First Line Treatment to EGFR Mutation Positive Advanced NSCLC With CNS Metastases
Brief Title: First Line Treatment in EGFR Mutation Positive Advanced NSCLC Patients With Central Nervous System (CNS) Metastases
Acronym: BM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alpha Biopharma (Jiangsu) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZD3759-003
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer; EGFR Gene Mutation; Brain Metastases
Keywords: Central Nervous System Metastases; Respiratory Tract Diseases; EGFR; Exon 19Del; L858R; Lung Neoplasm; Carcinoma, Non-Small-Cell Lung; Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Respiratory Tract Diseases; Lung Neoplasms; Neoplasms | interventions — AZD3759; Erlotinib Hydrochloride; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AZD3759 Group (Experimental): AZD3759 group will receive a 200 mg twice daily dose of AZD3759
  Interventions: Drug: AZD3759
- Erlotinib or Gefitinib Group (Active Comparator): SoC EGFR-TKI Erlotinib or Gefitinib Group will get EGFRTKI Erlotinib 150 mg or Gefitinib 250 mg PO Q.D
  Interventions: Drug: Erlotinib; Drug: Gefitinib

INTERVENTIONS:
Drug: AZD3759 — AZD3759 200mg PO BID.
  Arms: AZD3759 Group
Drug: Erlotinib — SoC EGFRTKI Erlotinib 150 mg PO Q.D
  Other Names: Tarceva
  Arms: Erlotinib or Gefitinib Group
Drug: Gefitinib — SoC EGFRTKI Gefitinib 250 mg PO Q.D
  Other Names: Iressa
  Arms: Erlotinib or Gefitinib Group

SUMMARY:
The first-line treatment with single agent AZD3759 results in superior Progression Free Survival (PFS) compared to Standard of Care (SoC) Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors (EGFR-TKI), in patients with advanced EGFR mutation positive non-small cell lung cancer (NSCLC) with Central Nervous System (CNS) metastasis

DETAILED DESCRIPTION:
This is a Phase II/III randomized, open-label, multicenter study to compare the efficacy and safety of first line single-agent AZD3759 vs. Erlotinib or Gefitinib treatment in patients with advanced EGFR mutation positive NSCLC with CNS metastases.

Eligible patients with documented EGFR mutation+ (L858R and/or Exon 19Del) TKI-naïve advanced NSCLC and documented intracranial disease will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Properly completed patient informed consent
2. Male or female aged at least 18 years
3. Histologically or cytologically confirmed diagnosis of NSCLC with activating EGFR mutations including L858R and/or Exon19Del. EGFR mutation status will be determined by local or central laboratory testing on tumour tissue or plasma utilizing a validated methodology which has been approved by the regulatory authority.
4. No prior treatment with chemotherapy, EGFR-TKIs, or biological therapies that are considered first line treatment for advanced NSCLC.
5. All patients must have a documented diagnosis of advanced (Stage IV) NSCLC with Magnetic Resonance Imaging (MRI) documented CNS metastases that include brain metastases (BM). BM + patients with co- existent leptomeningeal involvement are eligible for the study.
6. Eligible patients are not candidates for definitive surgical resection or radiation of all lesions in the opinion of the treating physician.
7. All patients must be stable without any systemic (oral or parenteral) corticosteroid or anticonvulsant therapy for at least 2 weeks prior to study treatment. Inhaled non-absorbable and topical corticosteroid use are permitted as indicated.
8. Patients may have prior placement of a properly functioning CNS shunt or Ommaya reservoir.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 with no deterioration over the previous 2 weeks.
10. Women of child-bearing potential and male subjects shall agree to take medically acceptable contraception measures while on study treatment and for 3 months following completion of study treatment. All women of child-bearing potential must have a negative blood pregnancy test at screening.
11. (a) For Patients with measurable CNS lesions must have AT LEAST ONE site of CNS lesion, which was not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter by MRI and which is suitable for accurate repeated measurements. Measurable extracranial disease is not required. (b) For Patients with non-measurable CNS lesions must have AT LEAST ONE extracranial lesion, which has not been previously irradiated, within the screening period that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) by CT/MRI and are suitable for accurate repeated measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
PFS assessed by Blinded Independent Central Radiological | 48 months
  To assess if first line treatment with AZD3759 results in significant PFS efficacy compared to Gefitinib or Erlotinib as determined by Blinded Independent Central Radiological (BICR) review using RECIST 1.1.

SECONDARY OUTCOMES:
PFS assess by investigator | 48 months
  Investigator assessment of PFS using RECIST 1.1
Intracranial PFS (iPFS) assessed by investigator | 48 months
  Intracranial PFS (iPFS) assessed by investigator using RECIST 1.1
Intracranial PFS (iPFS) assessed by BICR | 48 months
  Intracranial PFS (iPFS) assessed by Blinded Independent Central Radiological (BICR) using RECIST 1.1
Extracranial PFS (ePFS) assessed by investigator | 48 months
  Extracranial PFS (ePFS) assessed by investigator using RECIST 1.1
Extracranial PFS (ePFS) assessed by BICR | 48 months
  Extracranial PFS (ePFS) assessed by Blinded Independent Central Radiological (BICR) using RECIST 1.1
Objective Response Rate (ORR） assessed by investigator using RECIST 1.1 | 48 months
  Objective Response Rate (ORR) for Intracranial lesions and Extracranial lesions assessed separately by investigator using RECIST 1.1
Disease Control Rate (DCR) assessed by investigator using RECIST 1.1 | 48 months
  Disease Control Rate (DCR) for Intracranial lesions and Extracranial lesions assessed separately by investigator using RECIST 1.1
Duration of Response (DoR) assessed by investigator using RECIST 1.1 | 48 months
  Duration of Response (DoR) for Intracranial lesions and Extracranial lesions assessed separately by investigator using RECIST 1.1
Overall ORR assessed by investigator using RECIST 1.1 | 48 months
  Overall ORR assessed by investigator using RECIST 1.1
Overall DCR assessed by investigator using RECIST 1.1 | 48 months
  Overall DCR assessed by investigator using RECIST 1.1
Overall DoR assessed by investigator using RECIST 1.1 | 48 months
  Overall DoR assessed by investigator using RECIST 1.1
ORR for Intracranial lesions assessed by investigator using RANO-BM | 48 months
  ORR for Intracranial lesions assessed by investigator using RANO-BM
DCR for Intracranial lesions assessed by investigator using RANO-BM | 48 months
  DCR for Intracranial lesions assessed by investigator using RANO-BM
DoR for Intracranial lesions assessed by investigator using RANO-BM | 48 months
  DoR for Intracranial lesions assessed by investigator using RANO-BM
Overall Survival | 48 months
  Overall Survival
Change from baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30). | 48 months
  The 30-items questionnaire measures cancer patients' functioning and symptoms. The scale range of EORTC QLQ-C30 is 30-126. Lower values represent a better outcome.
Change from baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire BN20 (EORTC QLQ-BN20). | 48 months
  The 20-items questionnaire was used among brain cancer patients. The scale range of EORTC BN20 is 20-80. Lower values represent a better outcome.
Neurological function improvement rate assessed by Mini-Mental Status Examination (MMSE) | 48 months
  Neurological function improvement rate assessed by Mini-Mental Status Examination (MMSE)
Neurological function improvement rate assessed by RANO-BM criteria | 48 months
  Neurological function improvement rate assessed by RANO-BM criteria
Number of participants with treatment-related Adverse Events as assessed by CTCAE v5.0 | 48 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Number of participants with treatment-related Serious Adverse Events as assessed by CTCAE v5.0 | 48 months
  Number of participants with treatment-related Serious Adverse Events as assessed by CTCAE v5.0
Incidence of laboratory abnormalities collected by hematology tests during the study as assessed by CTCAE v5.0 | 48 months
  Incidence of laboratory abnormalities collected by hematology tests during the study as assessed by CTCAE v5.0
Incidence of laboratory abnormalities collected by biochemistry tests during the study as assessed by CTCAE v5.0 | 48 months
  Incidence of laboratory abnormalities collected by biochemistry tests during the study as assessed by CTCAE v5.0
Incidence of laboratory abnormalities collected byurinalysis tests during the study as assessed by CTCAE v5.0 | 48 months
  Incidence of laboratory abnormalities collected byurinalysis tests during the study as assessed by CTCAE v5.0
Rhythm, PR, R-R, QRS and QT intervals and an overall evaluation of ECG assessed during the study period. | 48 months
  Rhythm, PR, R-R, QRS and QT intervals and an overall evaluation of ECG assessed during the study period.
Systolic and Diastolic Blood Pressure assessed during the study period. | 48 months
  Systolic and Diastolic Blood Pressure assessed during the study period.
Pulse rate assessed during the study period. | 48 months
  Pulse rate to assessed during the study period.
Body temperature assessed during the study period. | 48 months
  Body temperature assessed during the study period.
PFS assess by BICR | 48 months
  Blinded Independent Central Radiological (BICR) assessment of PFS using modified RECIST 1.1.

OTHER OUTCOMES:
Pop-PK analysis | 48 months
  Population pharmacokinetic analysis
Exposure-Response analysis | 48 months
  explore the correlation in exposure and efficacy, exposure and safety in the Study

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, M.D., Study Chair — Guangdong Provincial People's Hospital; Myung-Ju Ahn, M.D., Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine; Jie Wang, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Qing Zhou, M.D., Principal Investigator — Guangdong Provincial People's Hospital
Locations (42):
- China (28):
  - China site, Hefei, Anhui
  - China site, Chongqing, China
  - China site, Fuzhou, Fujian
  - China site, Xiamen, Fujian
  - China site, Guangzhou, Guangdong
  - China site, Haerbin, Heilongjiang
  - China site, Zhengzhou, Henan
  - China site, Wuhan, Hubei
  - China site, Yichang, Hubei
  - China site, Changsha, Hunan
  - China site, Nanjing, Jiangsu
  - China site, Suzhou, Jiangsu
  - China site, Wuxi, Jiangsu
  - China site, Xuzhou, Jiangsu
  - China site, Yangzhou, Jiangsu
  - China site, Changchun, Jilin
  - China site, Xi'an, Shaanxi
  - China site 0123, Jinan, Shandong
  - China site, Linyi, Shandong
  - China site, Weifang, Shandong
  - China site, Yantai, Shandong
  - China site, Chengdu, Sichuan
  - China site, Kunming, Yunnan
  - China site, Hangzhou, Zhejiang
  - China site, Beijing
  - China site, Chongqing
  - China site, Shanghai
  - China site, Tianjin
- Singapore site, Singapore, Singapore
- South Korea (9):
  - Korea site, Daegu
  - Korea site, Gyeonggi-do
  - Korea site, Gyeongsang
  - Korea site, Incheon
  - Korea Site, Jungbuk
  - Korea Site, Seoul
  - Korea site, Seoul
  - Korea site, Suwon
  - Korea site, Ulsan
- Taiwan (4):
  - Taiwan site, Taichung
  - Taiwan site, Tainan
  - Taiwan site, Taipei
  - Taiwan site, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Q, Yu Y, Xing L, Cheng Y, Wang Y, Pan Y, Fan Y, Shi J, Zhang G, Cui J, Zhou J, Song Y, Zhuang W, Ma Z, Hu Y, Li G, Dong X, Feng J, Lu S, Wu J, Li J, Zhang L, Wang D, Xu X, Yang TY, Yang N, Guo Y, Zhao J, Yao Y, Zhong D, Xia B, Yang CT, Zhu B, Sun P, Shim BY, Chen Y, Wang Z, Ahn MJ, Wang J, Wu YL. First-line zorifertinib for EGFR-mutant non-small cell lung cancer with central nervous system metastases: The phase 3 EVEREST trial. Med. 2025 Jan 10;6(1):100513. doi: 10.1016/j.medj.2024.09.002. Epub 2024 Oct 9. PMID 39389055